CLINICAL TRIAL: NCT01670643
Title: The Effect of Video Camera Magnifier Use on Reading
Brief Title: Reading Performance With a Video Magnifier
Status: Completed | Type: Observational
Sponsor: Mary Lou Jackson (Other)
Responsible Party: Sponsor-Investigator, Mary Lou Jackson, Principal Investigator, Massachusetts Eye and Ear Infirmary
Organization: Massachusetts Eye and Ear Infirmary (Other)
Other Study IDs: 09-11-116; 09-11-116 (Other: Human Studies Committee MEEI)
Record Dates: First submitted 2010-12-06; First posted 2012-08-22 (Estimated); Last update posted 2017-03-27 (Actual); Status verified 2017-03

CONDITIONS: Macular Degeneration
Keywords: AMD; vision rehabilitation; video camera magnifier; IVI; DASS
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Video camera magnifier
  Interventions: Behavioral: Video camera magnifier

INTERVENTIONS:
Behavioral: Video camera magnifier — reading with video camera magnifier
  Other Names: Optelec video magnifier

SUMMARY:
The most common goal for patients with vision loss who present for vision rehabilitation is to be able to read. The video magnifier (a device which combines a video camera and a screen to view the print being magnified) is the device which most often allows low-vision individuals to read successfully for extended periods of time. Previous studies on the outcomes of vision rehabilitation have not identified which components of the vision rehabilitation are effective. The hypothesis of this project is that providing a video camera magnifier, with basic training in operating the device, will allow patients to enhance both objective reading ability and subjective report of reading competence.

DETAILED DESCRIPTION:
Patients will be given a video magnifier at initial consultation or at the end of vision rehabilitation

ELIGIBILITY:
Inclusion Criteria:

* Central field loss and decreased visual acuity in the better seeing eye (<20/40 & >20/400).
* New patient at MEEI Low Vision Rehabilitation Clinic

Exclusion Criteria:

* Dementia (Mini-Mental State Examination)
* Clinical depression (Geriatric Depression Scale)
* Patients who previously received vision rehabilitation
* Patients who have previously owned a desktop video magnifier

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2010-01; Primary Completion 2010-04 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Change in objective reading performance | baseline and one month
  The subject undergoes testing to determine the change in reading performance on an objective scale.

SECONDARY OUTCOMES:
Change in subjective reading performance | baseline and one month
  The subject is asked to describe subjectively how they feel their ability to read has either improved or decreased since using the reader.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Lou Jackson, MD, Principal Investigator — Vision Rehabilitation Center MEEI
Locations (1):
- Vision Rehabilitation Clinic Massachusetts Eye and Ear Infirmary, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No